CLINICAL TRIAL: NCT07222800
Title: AN INTERVENTIONAL, PHASE 3, DOUBLE-BLIND, RANDOMIZED STUDY TO EVALUATE THE EFFICACY AND SAFETY OF PF-08634404 IN COMBINATION WITH CHEMOTHERAPY VERSUS BEVACIZUMAB IN COMBINATION WITH CHEMOTHERAPY IN TREATMENT-NAÏVE PARTICIPANTS WITH METASTATIC COLORECTAL CANCER
Brief Title: A Study to Learn About the Study Medicine Called PF-08634404 in Combination With Chemotherapy in Adult Participants With Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C6461003; 2025-523521-18-00 (EU CTIS Number); Symbiotic-GI-03 (Other: Pfizer)
Record Dates: First submitted 2025-10-28; First posted 2025-10-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases; Colorectal Neoplasms
Keywords: mCRC; metastatic disease; first-line; metastatic colorectal cancer; colon cancer
MeSH Terms: conditions — Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases; Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms | interventions — Bevacizumab; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PF-08634404 + Chemotherapy (Experimental): Participants will receive PF-08634404 intravenously (IV) in combination with Chemotherapy.
  Interventions: Drug: PF-08634404; Drug: Chemotherapy
- Bevacizumab + Chemotherapy (Active Comparator): Participants will receive bevacizumab IV in combination with Chemotherapy.
  Interventions: Biological: Bevacizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: PF-08634404 — Solution for infusion
  Arms: PF-08634404 + Chemotherapy
Biological: Bevacizumab — Injection for intravenous use
  Other Names: Avastin
  Arms: Bevacizumab + Chemotherapy
Drug: Chemotherapy — Injection for intravenous use

SUMMARY:
The purpose of this study is to learn more about a new medicine called PF-08634404, and how well it works in people with cancer of the colon or rectum (CRC)). The goal is to understand if the new study medicine, combined with chemotherapy that is approved for colorectal cancer, can help people whose cancer has spread or returned after treatments taken before.

To join the study, participants must meet the following conditions:

* Be 18 years or older.
* Have colorectal cancer that has spread to other parts of your body.
* Be in good enough health to receive study treatment.
* Should not be pregnant before starting treatment.

Participants will be randomized (like flipping a coin) to one of 2 different treatment arms. The first arm (Arm A) will include the new medicine PF-08634404 in combination with chemotherapy that is approved for colorectal cancer, and the second arm (Arm B) will include an approved medicine for colorectal cancer, called Bevacizumab, in combination with chemotherapy that is approved for this type of cancer. Participants and their doctors will not know which arm they are being assigned to. Participants will receive all the study medications through intravenous (IV) infusions, which means the medicine is given directly into a vein. The treatment will be given in cycles, and participants may continue receiving it if it is helping and they are not experiencing serious side effects.

The medicine will be given at a clinical site, where trained medical staff will check participants during and after each treatment.

* The study is expected to last approximately 33 months for each participant.
* Participants will have regular visits to the study site for treatment, health checks, and tests.
* After stopping treatment, participants will return for a final visit about 30 to37 days later to check their health and review any side effects.
* Follow-up will continue every 12 weeks by phone or in person or by reviewing health records to check on health status and any new treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed colorectal adenocarcinoma.
* Evidence of Stage IV metastatic disease.
* No prior systemic therapy for metastatic disease.
* Eastern Cooperative Oncology Group performance status (ECOG) 0-1
* At least one measurable lesion according to RECIST 1.1 per Investigator assessment.
* Adequate hepatic, liver, and renal function

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Locally confirmed BRAF V600E mutation
* Locally confirmed microsatellite instability (MSI)-high or DNA mismatch repair deficiency (dMMR) colorectal cancer
* Participants with known active symptomatic CNS lesions, including leptomeningeal metastasis, brainstem, meningeal, or spinal cord metastases or compression
* Clinically significant risk of hemorrhage or fistula
* Major surgery or severe trauma within 4 weeks prior to the first dose, or planned major surgery during the study
* History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation
* Any Grade ≥3 bleeding/hemorrhage events within 28 days of Cycle 1 Day 1, or prior history of clinically significant bleeding events
* Clinically significant cardiovascular disease, or other comorbidities, within 6 months prior to first dose
* Participants with active autoimmune diseases requiring systemic treatment within the past 2 years
* Evidence of non-infectious or drug-induced interstitial lung disease (ILD) pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2030-03-29 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) by Blinded Independent Central Review (BICR) | Approximately 4 years
  Progression-free survival is defined as the time from the date of randomization to the date of the first documentation of objective progressive disease (PD) assessed by BICR per RECIST 1.1, or death due to any cause, whichever occurs first.
Overall survival (OS) | Approximately 4 years
  Overall survival defined as the time from the date of randomization to the date of death due to any cause.

SECONDARY OUTCOMES:
PFS per RECIST 1.1 by investigator assessment | Approximately 4 years
  Progression Free Survival (PFS) is defined as the time from the date of randomization to the date of the first documentation of objective PD assessed by investigator per RECIST 1.1, or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) by BICR | Approximately 4 years
  The proportion of participants who have a confirmed CR or PR, as best overall response assessed by BICR as per RECIST 1.1.
Objective Response Rate (ORR) by investigator | Approximately 4 years
  The proportion of participants who have a confirmed CR or PR, as best overall response assessed by investigator as per RECIST 1.1.
Duration of Response (DOR) by BICR | Approximately 4 years
  The time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the date of the first documentation of PD as determined by BICR assessment per RECIST 1.1, or death due to any cause, whichever occurs first.
DOR by investigator | Approximately 4 years
  The time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the date of the first documentation of PD as determined by Investigator per RECIST 1.1, or death due to any cause, whichever occurs first.
PFS2 (PFS after next-line therapy) by investigator | Approximately 4 years
  PFS2 is defined as the time from the date of randomization to the date of second objective disease progression or death due to any cause, whichever occurs first. Second objective disease progression is PD after the start of subsequent anticancer therapy (excluding curative surgery) as assessed by the investigator.
Number of Participants with Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Through 90 days after the last study intervention; Approximately 4 years
Number of Participants With Clinical Laboratory Abnormalities | Through 90 days after the last study intervention; Approximately 4 years
Pharmacokinetics (PK): Serum concentration of PF-08634404 | Approximately 21 months
Immunogenicity: Incidence of positive Anti-Drug Antibody (ADA) | Approximately 21 months
  To characterize the immunogenicity of PF-08634404
Mean scores and Change from baseline in the global health status/quality of life (QoL) score on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Approximately 4 years
  The EORTC QLQ-C30 is a questionnaire for quantitative measure of health-related quality of life pertinent to participants with a broad range of cancers who are participating in international clinical trials.
Mean score change from baseline in participant reported function and symptoms scales per EORTC QLQ-CR29 | Approximately 4 years
  The EORTC QLQ-CR29 is a supplemental colorectal cancer-specific module with measures of symptoms associated with colorectal cancer.
Time to definitive deterioration (TTdD) in the global health status/QoL score on the EORTC QLQ-C30 | Approximately 4 years
  TTdD is defined as the time from date of randomization to first onset of Patient Reported Outcome (PRO) deterioration without subsequent recovery.
Time to definitive deterioration (TTdD) in participant reported function and symptoms per EORTC QLQ-CR29 | Approximately 4 years
  TTdD is defined as the time from date of randomization to first onset of Patient Reported Outcome (PRO) deterioration without subsequent recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (8):
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Cancer Care Centers of Brevard, Inc., Palm Bay, Florida
  - Illinois Cancer Care, Canton, Illinois
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Oncology Associates of Oregon, P.C., Albany, Oregon
  - Texas Oncology - West Texas, Odessa, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
- Australia (2):
  - Icon Cancer Centre Wesley, Auchenflower
  - Icon Cancer Centre Hobart, Hobart
- Japan (5):
  - Kyushu University Hospital, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka
  - National Hospital Organization Osaka Medical Center, Osaka
  - Saitama Prefectural Cancer Center, Saitama
  - The Cancer Institute Hospital of JFCR, Tokyo
- Pan American Center for Oncology Trials, LLC, Rio Piedras, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C6461003